CLINICAL TRIAL: NCT06027879
Title: Anti-viral T-cell Therapy by Gamma Capture for High-risk Patients With Acquired or Inherited Immune Defects
Brief Title: Anti-viral T-cell Therapy by Gamma Capture
Acronym: Gamma Capture
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Paul Szabolcs (Other)
Responsible Party: Sponsor-Investigator, Paul Szabolcs, Chief, Division of Blood and Marrow Transplantation and Cellular Therapies, Medical Director of the Stem Cell Laboratory, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23030062
Record Dates: First submitted 2023-07-05; First posted 2023-09-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Adenovirus; Cytomegalovirus Infections; Epstein-Barr Virus Infections
MeSH Terms: conditions — Adenoviridae Infections; Cytomegalovirus Infections; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Viral Specific T-Lymphocytes (Experimental): Viral Specific T-Lymphocytes Peripheral blood mononuclear cells will be collected from the donor and loaded onto our Miltenyi Biotec CliniMACS Prodigy® or CliniMACS® Plus where they will be stimulated in vitro with viral-specific antigen(s). The cells are then immunomagnetically labeled with interferon gamma via the cytokine capture system. By this method, viral specific, gamma-secreting T cells, are captured in a closed, sterile system.
  Interventions: Biological: Specific T- Lymphocytes

INTERVENTIONS:
Biological: Specific T- Lymphocytes — Peripheral blood mononuclear cells will be collected from the donor and loaded onto Miltenyi Biotec CliniMACS Prodigy® or CliniMACS® Plus where they will be stimulated in vitro with Adenovirus viral-specific antigen(s). The cells are then immunomagnetically labeled with interferon gamma via the cytokine capture system, captured and infused.

SUMMARY:
The primary purpose of this phase I/II study is to evaluate whether partially matched, ≥1/6 Human Leukocyte Antigens (HLA) -matched, viral specific T cells have efficacy against adenovirus, Cytomegalovirus (CMV), and Epstein Barr Virus (EBV) in subjects who have previously received any type of allogeneic Hematopoietic Cell transplant (HCT) or solid organ transplant (SOT) or have compromised immunity. Reconstitution of anti-viral immunity by donor-derived cytotoxic T lymphocytes has shown promise in preventing and treating infections with adenovirus, CMV, and EBV. However, the weeks taken to prepare patient-specific products, and cost associated with products that may not be used limits their value. This trial will evaluate viral specific T cells generated by gamma capture technology. Eligible patients will include HCT and/or SOT recipients, and/or patients with compromised immunity who have adenovirus, CMV, or EBV infection or refractory viremia that is persistent despite standard therapy. Infusion of the cellular product will be assessed for safety and efficacy.

DETAILED DESCRIPTION:
Enrollment for existing UPMC patients.

Ideally, subjects will receive up to ≤1 x 105 (100,000) viable CD3 cells/kg however actual cell dose of infusion will be based upon available cells and subject's clinical picture. Historically, subjects have received all available cells after the gamma capture procedure.

Two-weeks post initial cellular infusion, subject may be eligible to receive additional cellular infusions. If so, either the same or an alternative donor may be considered however, a subject will not receive more than 3 infusions from one donor or exceed 6 infusions in total from all donors. Infusions will be a minimum of 14-days apart. Subjects will not receive additional infusions if they exhibit Graft Versus Host Disease (GvHD) or Cytokine Release Syndrome (CRS) Grade II or higher, according to CTCAE v5.

If a subject is to receive a second infusion, eligibility and baseline data collection will not be repeated for the recipient or original donor, unless necessary per institutional guidelines. Should an alternative donor be selected for an infusion, eligibility of the new donor will need confirmed. Pregnant donors may be considered if medically suitable.

Two weeks post-initial cellular infusion, the following criteria will be assessed to determine if additional infusions are necessary:

* Complete response: Return to normal range as defined by specific assay used and clinical signs and symptoms. These subjects are not eligible to receive an additional cellular infusion.
* Partial response: Decrease in viral load of at least 50% from baseline or significant improvement of clinical signs. The clinical response is further defined as meeting one or more of the following criteria and no worsening in any of the others:

  1. Absence of fever, if fever is present at baseline
  2. No need for pressors, if on pressors at baseline
  3. No need for oxygen and/or mechanical ventilation, if needed at baseline
  4. Decrease in stool output, if is diarrhea present at baseline

These subjects may receive additional cellular infusions as clinically indicated:

* Stable disease: Changes insufficient to qualify as partial response or progression. These subjects are eligible to receive additional cellular infusions.
* Progression: Increase in viral load of at least 50% from baseline or dissemination to other sites of disease. These subjects are eligible to receive additional cellular infusions.

Subjects are followed for six months post initial viral-specific T cell infusion. If a subject receives additional infusions, GVHD and adverse events only will be followed for a minimum of three months from last infusion, even if extending beyond the six-month follow-up from the first infusion. Data may be abstracted from subjects' medical charts for an additional 1 year after most recent viral-specific T cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patient, parent, or legal guardian must have given written informed consent, according to FDA guidelines. For pediatric subject who are developmentally able, assent or affirmation will be obtained, if feasible.
2. Male or female, 1 month through 75 years old, inclusive, at the time of informed consent.
3. Prior allogeneic hematopoietic stem cell transplant (bone marrow, peripheral blood stem cells, single or double cord blood), OR prior solid organ transplant (liver, kidney, lung and/or heart, intestinal, or multivisceral), OR diagnosis of primary immunodeficiency OR current/recent administration of immunosuppressive therapy for cancer or autoimmune disease.
4. Negative pregnancy test for females ≥10 years old or who have reached menarche, unless surgically sterilized. All females of childbearing potential and lactation must agree to use an FDA approved method of birth control for the duration of their participation.
5. Clinical status, at the time of consent, amendable to tapering of steroids to less than 1 mg/kg/day prednisone (or equivalent) prior to cellular infusion.
6. Diagnosis of Adenovirus, CMV, or EBV infection, persistent despite standard therapy.

A. Adenovirus Infection or Disease:

1. Active adenovirus infection: (i.e. gastroenteritis, pneumonia, hemorrhagic cystitis, hepatitis, pancreatitis, meningitis) defined as the demonstration of adenovirus by biopsy specimen from affected site(s) (by culture or histology), or the detection of adenovirus by culture, PCR or direct fluorescent antibody stain in fluid in the presence of worsening or persistent clinical or imaging findings despite at least 14 days of appropriate antiviral therapy (i.e. cidofovir, brincidofovir, or other available pharmacological agents) OR
2. Refractory adenoviremia: defined as DNAemia >5000 copies/mL or <1 log decrease after at least 2 weeks of appropriate antiviral therapy (i.e. cidofovir, brincidofovir, or other available pharmacological agents) OR
3. Intolerance of or contraindication to antiviral medications.

B.CMV Infection or Disease:

1. Active CMV infection: (i.e. pneumonia, meningitis, retinitis, hepatitis, hemorrhagic cystitis, and/or gastroenteritis) defined as the demonstration of CMV by biopsy specimen from affected site(s) (by culture or histology) or the detection of CMV by culture, PCR or direct fluorescent antibody stain in fluid in the presence of worsening or persistent clinical or imaging findings despite at least 14 days of appropriate antiviral therapy (i.e. Foscarnet, ganciclovir, cidofovir, or other available pharmacological agents) OR
2. Refractory CMV viremia: defined as the continued presence of DNAemia, with ≥2,000 IU/mL or <1 log decrease after at least 14 days of appropriate antiviral therapy (i.e. Foscarnet, ganciclovir, cidofovir, or other available pharmacological agents) OR
3. Intolerance of or contraindication to antiviral medications.

C. EBV Infection or Disease:

1. Biopsy proven lymphoma or posttransplant lymphoproliferative disease with EBV genomes detected in tumor cells by immunocytochemistry (i.e. EBER positive) or in situ PCR, OR
2. Clinical or imaging findings consistent with EBV lymphoma and associated elevated EBV viral load in peripheral blood in a patient where biopsy is deemed too high risk, OR
3. Failure of antiviral therapy, as determined by one of the two bullets below after three weeks of anti-CD20 targeted therapy such as Rituximab.

i. There was an increase or less than 50% response at sites of lymphoma disease or lymphoproliferation.

ii. There was a rise or a fall of less than 50% in EBV viral load in peripheral blood of PTLD patients.

Exclusion Criteria:

1. Received Antithymocyte Globulin (ATG) or Alemtuzumab within 28 days of viral-specific T cell infusion and a lack of evidence of T cell survival, defined by <10 CD3+ T cells/uL (in unique situations, plasmapheresis may be considered).
2. Active acute GVHD grades II-IV.
3. Received donor lymphocyte infusion, with the exception of a fraction of an umbilical cord blood, within 14 days of viral-specific T cell infusion. Subjects receiving a fraction of an umbilical cord blood within 14 days of the viral-specific T cell infusion will not be excluded.
4. Active and uncontrolled relapse of malignancy (other than EBV+ post-transplant lymphoproliferative disorder or lymphoma).
5. Received an investigational product in the preceding 2 weeks (prior to infusion) that may impact Viral Specific T-cells (VST) survival.
6. Females of child bearing potential must not be lactating.
7. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks to participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Grade III-IV Acute GvHD | Day 0
  The number of patients who develop Grade III-IV acute graft versus host disease (GVHD) attributed to the viral specific T cells.
Grade III-IV Acute GvHD | 1 month from first cellular infusion
  The number of patients who develop Grade III-IV acute graft versus host disease (GVHD) attributed to the viral specific T cells.
Grade III-IV Acute GvHD | 3 month from first cellular infusion
  The number of patients who develop Grade III-IV acute graft versus host disease (GVHD) attributed to the viral specific T cells.
Grade III-IV Acute GvHD | 6 month from first cellular infusion
  The number of patients who develop Grade III-IV acute graft versus host disease (GVHD) attributed to the viral specific T cells.
Clinical response to treatment of viral infection | 1 month from first cellular infusion
  Rate of Elimination or reduction of oxygen dependence identified at baseline
Clinical response to treatment of viral infection | 1 month from first cellular infusion
  Rate of Resolution of diarrhea attributable to the viral disease, less than 4 stools daily
Clinical response to treatment of viral infection | 1 month from first cellular infusion
  Rate of Resolution of fever, attributable to viral disease
Clinical response to treatment of viral infection | 1 month from first cellular infusion
  Rate of Resolution or improvement of radiographic findings attributable to viral disease
Clinical response to treatment of viral infection | 1 month from first cellular infusion
  Rate of Resolution or improvement of lymphadenopathy attributable to EBV, and ophthalmic findings attributable to CMV retinitis
Clinical response to treatment of viral infection | 3 month from first cellular infusion
  Rate of Elimination or reduction of oxygen dependence identified at baseline
Clinical response to treatment of viral infection | 3 month from first cellular infusion
  Rate of Resolution of diarrhea attributable to the viral disease, less than 4 stools daily
Clinical response to treatment of viral infection | 3 month from first cellular infusion
  Rate of Resolution of fever, attributable to viral disease
Clinical response to treatment of viral infection | 3 month from first cellular infusion
  Rate of Resolution or improvement of radiographic findings attributable to viral disease
Clinical response to treatment of viral infection | 3 month from first cellular infusion
  Rate of Resolution or improvement of lymphadenopathy attributable to EBV, and ophthalmic findings attributable to CMV retinitis
Clinical response to treatment of viral infection | 6 months from first cellular infusion
  Rate of Elimination or reduction of oxygen dependence identified at baseline
Clinical response to treatment of viral infection | 6 months from first cellular infusion
  Rate of Resolution of diarrhea attributable to the viral disease, less than 4 stools daily
Clinical response to treatment of viral infection | 6 months from first cellular infusion
  Rate of Resolution of fever, attributable to viral disease
Clinical response to treatment of viral infection | 6 months from first cellular infusion
  Rate of Resolution or improvement of radiographic findings attributable to viral disease
Clinical response to treatment of viral infection | 6 months from first cellular infusion
  Rate of Resolution or improvement of lymphadenopathy attributable to EBV, and ophthalmic findings attributable to CMV retinitis

SECONDARY OUTCOMES:
1-year overall survival from first cellular infusion (continuous) | First cellular infusion to 1 year post first cellular infusion
  Number of deaths that occurred from treatment
Incidence of Graft rejection | 3 months after last cellular infusion
  How frequent, if any, graft rejection occurs
Incidence of Graft rejection | 6 months after last cellular infusion
  How frequent, if any, graft rejection occurs
Incidence of Mechanical ventilation exceeding 48 hours | 3 months after last cellular infusion
  How long, if any
Incidence of Mechanical ventilation exceeding 48 hours | 6 months after last cellular infusion
  How long, if any
Usage of concomitant antiviral agents | First cellular infusion to 1 year post first cellular infusion
  The introduction of concomitant antiviral medication post infusion, if any
Immune reconstitution with focus on adaptive T cell immunity and viral-specific responses | 1 month following first cellular infusion
  The pace of systemic immune reconstitution, measured by the increased number of CD4+ T lymphocytes.
Immune reconstitution with focus on adaptive T cell immunity and viral-specific responses | 3 months following first cellular infusion
  The pace of systemic immune reconstitution, measured by the increased number of CD4+ T lymphocytes.
Incidence of severe or extensive chronic GVHD | 6 months from first cellular infusion
  The number of patients who develop chronic graft versus host disease (GVHD) post first infusion based on Clinical Chronic GvHD Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Paul Szabolcs, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No